CLINICAL TRIAL: NCT01953029
Title: Mechanisms of Myocardial Infarction in Women With Non Obstructive Coronary Artery Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Miry Blich MD, Senior Cardiologist, Rambam Health Care Campus
Other Study IDs: 0541-12-RMB
Record Dates: First submitted 2013-09-23; First posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- non obstructive coronary disease: non obstructive coronary disease
  Interventions: Procedure: cardiac imajing

INTERVENTIONS:
Procedure: cardiac imajing — Cardiac MRI

SUMMARY:
The objective of our work to determine the mechanisms of myocardial infarction in women without obstructive coronary artery disease.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death for women. Acute coronary syndrome (ACS) is usually characterized by a sudden erosion of the endothelial wall or rupture of a plaque.However, women with ACS are less likely than men to have either classic symptoms or obstructive coronary artery disease but paradoxically have a worse prognosis. Different data from the literature indicate that there may be different pathophysiological mechanisms, afflicting men and women somewhat differently.Between 5% and 30% of patients with ACS undergoing coronary angiography are found to have non visible or non obstructive coronary disease (NOCD). This is 2-3 times more common in women than in men. Several pathogenetic mechanism of myocardial infarction (MI) in the absence of obstructive coronary artery disease (OCD) have been postulated, including among others atherosclerosis with plaque disruption that does not lead to luminal occlusion ,endothelial dysfunction, vasospasm , distal microembolization and microvascular dysfunction. However the data are extremely limited.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old, not pregnant
* with acute non ST elevation myocardial infarction (admitted within 12 hours from beginning of symptoms)
* who are candidates for coronary arteriography during the hospitalization. -

Exclusion Criteria:

*Women with troponin elevation caused by other causes -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
MORTALITY | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: Miry Blich, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Heath Care Campus, Haifa, Israel